CLINICAL TRIAL: NCT06281431
Title: A Comparative Effect of Echogenic Needle for Nerve Block on Acute and Chronic Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPSP
Record Dates: First submitted 2024-01-14; First posted 2024-02-28 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Chronic Postoperative Pain
Keywords: Visualized nerve block needle; Acute pain; Chronic pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Echogenic nerve block needle (Experimental): Using a echogenic nerve block needle.
  Interventions: Procedure: Echogenic nerve block needle
- Non-echogenic nerve block needle (Other): Using a common nerve block needle.
  Interventions: Procedure: Non-echogenic nerve block needle

INTERVENTIONS:
Procedure: Echogenic nerve block needle — A 22G 8-cm echogenic nerve block needle (LEAPMED, CHINA) is selected for the procedure, administered under ultrasound guidance. Subsequently, a volume of 20 ml 0.375% ropivacaine is injected at the needle's tip for analgesic effect. The spread of the medication will be assessed through short- and long-axis imaging perspectives. Following this, evaluations are conducted to assess acute postoperative pain as well as chronic postoperative pain. Parameters such as the duration of nerve blockade, the incidence of punctures, and any associated complications are all meticulously appraised.
  Arms: Echogenic nerve block needle
Procedure: Non-echogenic nerve block needle — A 22G 8-cm thin wall low bottom nerve block needle (KDL, CHINA) is selected for the procedure, administered under ultrasound guidance. Subsequently, a volume of 20 ml 0.375% ropivacaine is injected at the needle's tip for analgesic effect. The distribution of the medication will be assessed using short- and long-axis imaging perspectives. Following this, evaluations are conducted to assess acute postoperative pain as well as chronic postoperative pain. Parameters such as the duration of nerve blockade, the number of punctures, and any associated complications are all meticulously appraised.
  Arms: Non-echogenic nerve block needle

SUMMARY:
Surgical pain is a common complication after surgery, affecting patient recovery and treatment quality. >20% of patients suffer from chronic postoperative pain. China has >70 million surgeries yearly. Nerve block manages postoperative pain, with developing nerve block needles now used in clinics. Developed needles may have better pain management effects than non-developed ones, but their effect on reducing chronic pain remains unclear. This study aims to explore the effect of developed nerve block needles on postoperative pain and compare them to non-developed needles, providing new ideas and methods for pain management.

DETAILED DESCRIPTION:
Surgical pain is one of the common complications after surgery, which seriously affects the recovery and treatment quality of patients. More than 20% of patients will suffer from postoperative chronic pain. According to the data of the National Bureau of Statistics, there are more than 70 million surgeries in China every year. Nerve block is one of the most commonly used methods for postoperative pain management in clinical practice. In recent years, the developing nerve block needle has gradually begun to be used in clinical practice. Compared with the ordinary non-developing nerve block needle, it may have a better effect on pain management after surgery, but whether it has a reduction effect on chronic pain after surgery is still unknown. The purpose of this study is to explore the effect of developing nerve block needle on postoperative pain, and to compare the difference between it and the common non-developing nerve block needle, so as to provide new ideas and methods for postoperative pain management.

ELIGIBILITY:
Inclusion Criteria:

1. The age is above 18 years old and below 70 years old.
2. patients whose surgical sites were in the chest, abdomen, upper limbs or lower limbs, including lobectomy, cholecystectomy, gastrointestinal resection, hysterectomy and other elective operations.
3. This operation was the first operation during the hospitalization.
4. Consent to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Patients with a history of alcohol or drug addiction.
2. Patients with disturbance of consciousness before operation.
3. Other conditions considered by the attending physician or researcher to be inappropriate for the study;
4. History of chronic pain.
5. Abnormal coagulation function.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Chronic postoperative pain | The third month after surgery.
  Incidence of Chronic pain assessment from 3 months after surgery
Moderate to severe pain | from end of surgery to 24 hours after surgery.
  Pain intensity (assessed by number rating scale, 0 represents no pain, 10 represents intolerable pain) more than 4

SECONDARY OUTCOMES:
Acute postoperative pain | From the ending of surgery to leaving the postanesthesia care unit, an average of 30 minutes
  Pain intensity (assessed by number rating scale, 0 represents no pain, 10 represents intolerable pain) more than 4
Acute postoperative pain | From return to the ward to 12 hours after return to the ward
  Pain intensity (assessed by number rating scale, 0 represents no pain, 10 represents intolerable pain) more than 4
Acute postoperative pain | From 12 hours after return to the ward to 24 hours after return to the ward
  Pain intensity (assessed by number rating scale, 0 represents no pain, 10 represents intolerable pain) more than 4
Puncture operation time | From the ending of surgery to leaving the postanesthesia care unit, an average of 30 minutes
  Time from needle insertion to needle extraction
Number of needle passes | From the ending of surgery to leaving the postanesthesia care unit, an average of 30 minutes
  The number of times the needle is withdrawn more than 2 cm and resited

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, ph.D, Study Chair — The Second Affiliated Hospital, Chongqing Medical University
Locations (1):
- He Huang, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within one year